CLINICAL TRIAL: NCT03270059
Title: The Feasibility of Steady State CBV Mapping Using Ferumoxytol Immediately After Gadolinium Enhanced MRI of the CNS
Brief Title: Gadolinium and Ferumoxytol MRI in Diagnosing Patients With Abnormalities in the Central Nervous System
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Celgene Corporation (Industry); Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Michael F. Regner, M.D., M.S., Principal Investigator, OHSU Knight Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY00017028; NCI-2017-01460 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00017028 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2017-08-30; First posted 2017-09-01 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Central Nervous System Neoplasm; Cranial Nerve Disorder; Metastatic Malignant Neoplasm in the Brain
MeSH Terms: conditions — Central Nervous System Neoplasms; Cranial Nerve Diseases; Brain Neoplasms | interventions — Ferrosoferric Oxide; Gadolinium; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I (gadolinium, ferumoxytol, MRI) (Experimental): Patients receive gadolinium IV and then ferumoxytol IV and undergo MRI over 60 minutes on day 1.
  Interventions: Drug: Ferumoxytol; Drug: Gadolinium; Procedure: Magnetic Resonance Imaging
- Group II (ferumoxytol, gadolinium, MRI) (Experimental): Patients receive ferumoxytol IV and then gadolinium IV and undergo MRI over 60 minutes on day 1.
  Interventions: Drug: Ferumoxytol; Drug: Gadolinium; Procedure: Magnetic Resonance Imaging

INTERVENTIONS:
Drug: Ferumoxytol — Given IV
  Other Names: Feraheme; Ferumoxytol Non-Stoichiometric Magnetite
Drug: Gadolinium — Given IV
  Other Names: Gd
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging

SUMMARY:
This phase II trial studies how well gadolinium and ferumoxytol magnetic resonance imaging (MRI) work in diagnosing patients with abnormalities in the central nervous system. Diagnostic procedures, such as gadolinium and ferumoxytol MRI, may help find and diagnose abnormalities in the central nervous system.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To test if prior gadolinium administration affects vascular imaging using ferumoxytol.

II. To test signal changes of T2*w multi-echo fast field echo (mFFE) scans before and after contrast agent injection.

SECONDARY OBJECTIVES:

I. To test if ferumoxytol affects gadolinium enhanced MRI. II. To test if steady state cerebral blood volume (CBV) maps are different at various magnetic field strengths.

EXPLORATORY OBJECTIVES:

I. To explore late ferumoxytol enhancement (optional MRI) hours to days after ferumoxytol administration in various brain pathologies.

II. To evaluate the effects of ferumoxytol on malignant and non-malignant lesions in head & neck, and liver lesions

OUTLINE: Patients are randomized into 1 of 2 groups.

GROUP I: Patients receive gadolinium intravenously (IV) and then ferumoxytol IV and undergo MRI over 60 minutes on day 1.

GROUP II: Patients receive ferumoxytol IV and then gadolinium IV and undergo MRI over 60 minutes on day 1.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have one of the following:

  * Neurological findings (i.e. headache, loss of consciousness, paresis, cranial neuropathy, seizures, etc.)
  * Radiological abnormalities in the brain (neoplastic or non-neoplastic in nature)
  * Neoplastic process elsewhere in the body that may affect the brain (i.e. possible metastasis, vascular compromise, treatment related changes, etc.)
* Subjects must be able to undergo MRI imaging without anesthesia
* Subjects must be at least 10 years of age
* All subjects, or their legal guardians, must sign a written informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization in accordance with institutional guidelines
* Sexually active women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; surgical intervention i.e. tubal ligation or vasectomy; post-menopausal < 6 months; or abstinence) for at least two months after each cycle of the study; should a female become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately

Exclusion Criteria:

* Subjects with clinically significant signs of uncal herniation, such as acute pupillary enlargement, rapidly developing motor changes (over hours), or rapidly decreasing level of consciousness, are not eligible
* Subjects with known allergic or hypersensitivity reactions to parenteral iron, parenteral dextran, parenteral iron-dextran, or parenteral iron-polysaccharide preparations (Ferumoxytol Investigator's Drug Brochure, 2009); subjects with significant drug or other allergies or autoimmune diseases may be enrolled at the investigator's discretion
* Subjects who are pregnant or lactating or who suspect they might be pregnant
* Subjects who have a contraindication for MRI: metal in their bodies (a cardiac pacemaker or other incompatible device), are severely agitated, or have an allergy to gadolinium containing contrast material
* Subjects with known iron overload (genetic hemochromatosis); in subjects with a family history of hemochromatosis, hemochromatosis must be ruled out prior to study entry with normal values of the following blood tests: transferrin saturation (TS) test and serum ferritin (SF) test; all associated costs will be paid by the study
* Subject who have received ferumoxytol within 3 weeks of study entry
* Subjects with three or more drug allergies from separate drug classes

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2017-10-06 (Actual); Primary Completion 2026-08-15 (Estimated); Study Completion 2027-08-15 (Estimated)

PRIMARY OUTCOMES:
Visualization of normal vasculature | Up to 5 years
  Primary analysis will use the average score of the two readers. The mean difference and the associated 95% confidence interval (CI) between the two groups will be estimated using a linear regression model. Equivalence will be claimed if the 95% CI does not include 0.4 on either side (equivalence margin is 0.4).
Visualization of abnormal vasculature | Up to 5 years
  Primary analysis will use the average score of the two readers. The mean difference and the associated 95% CI between the two groups will be estimated using a linear regression model. Equivalence will be claimed if the 95% CI does not include 0.4 on either side (equivalence margin is 0.4).
Visualization of normal anatomical structures | Up to 5 years
  Primary analysis will use the average score of the two readers. The mean difference and the associated 95% CI between the two groups will be estimated using a linear regression model. Equivalence will be claimed if the 95% CI does not include 0.4 on either side (equivalence margin is 0.4).
Identification of the lesion corresponding areas on cerebral blood volume (CBV) maps | Up to 5 years
  Will assess the confidence in identifying the lesion corresponding areas on CBV maps as well as signal change (deltaR2*) and relative cerebral blood volume. Primary analysis will use the average score of the two readers. The mean difference and the associated 95% CI between the two groups will be estimated using a linear regression model. Equivalence will be claimed if the 95% CI does not include 0.4 on either side (equivalence margin is 0.4).

SECONDARY OUTCOMES:
Contrast enhancement | Up to 5 years
  The mean difference and the associated 95% CI before versus after ferumoxytol in the three visualization variables will be estimated using a paired t-test based on the average score of the two readers. Will use the same equivalence margin of 0.4. To compare the two magnetic field strengths, will also use a linear regression model to analyze contrast to noise ratios, Image homogeneity and susceptibility artifacts (the latter two based on average score of the two readers).
Border delineation | Up to 5 years
  The mean difference and the associated 95% CI before versus after ferumoxytol in the three visualization variables will be estimated using a paired t-test based on the average score of the two readers. Will use the same equivalence margin of 0.4. To compare the two magnetic field strengths, will also use a linear regression model to analyze contrast to noise ratios, Image homogeneity and susceptibility artifacts (the latter two based on average score of the two readers).
Internal morphology | Up to 5 years
  The mean difference and the associated 95% CI before versus after ferumoxytol in the three visualization variables will be estimated using a paired t-test based on the average score of the two readers. Will use the same equivalence margin of 0.4. To compare the two magnetic field strengths, will also use a linear regression model to analyze contrast to noise ratios, Image homogeneity and susceptibility artifacts (the latter two based on average score of the two readers).

CONTACTS AND LOCATIONS:
Overall Officials: Michael F Regner, MD, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States